CLINICAL TRIAL: NCT03427385
Title: Minimum Effective Local Anesthetic Dose for Adductor Canal Block for Knee Analgesia - a Preliminary Study
Brief Title: Minimum Local Anesthetic Dose for Adductor Canal Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 11-0635-A
Record Dates: First submitted 2018-01-26; First posted 2018-02-09 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Neuromuscular Blockade
Keywords: Neuromuscular blockade
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Minimum Effective dose (Experimental): Local anesthetic Ropivacaine 0.5% injection for adductor canal block
  Interventions: Drug: Ropivacaine 0.5%

INTERVENTIONS:
Drug: Ropivacaine 0.5% — The volume of local anesthetic Ropivacaine 0.5% will be determined by the response (success or failure of block, 30 minutes after local anesthetic injection) of the previous patient in that group. Block success is defined as an absence of ice sensation in the knee within 30 min of ropivacaine administration accompanied by tolerance to tetanic electrical stimulation (TES) at 60 mA(milliamp) for 5 seconds.
  Other Names: Naropin

SUMMARY:
The purpose of this study is to determine the minimum dose of ropivacaine 0.5%, required to produce pain relief without weakening the leg muscles.

DETAILED DESCRIPTION:
The post-operative period after a Total Knee Arthroplasty (TKA) is known to be especially painful for the first 24 hours. Significant pain can persist up to 3 days in some cases. Successful management of pain post TKA is therefore regarded as essential to early recovery, rehabilitation and timely discharge.

Until now, multiple modes of analgesia have been employed including intravenous patient-controlled analgesia, continuous femoral nerve block and epidural analgesia. These are all effective alternatives but each is limited by side effects. Epidural analgesia provides excellent pain control and has been associated with early rehabilitation despite its negative impact on ambulation in the immediate peri-operative period. Additionally, an increased risk of spinal hematoma has been reported with epidural analgesia and peri-operative low molecular weight heparin prophylaxis. For this reason, epidural analgesia is not routinely offered to patients undergoing TKA today.

A multimodal analgesic approach centered on the use of continuous femoral nerve blocks has been more recently favoured, providing superior analgesia and less opioid-related side effects than a systemic opioid-based regimen. However, femoral nerve blockade is also associated with significant quadriceps muscle weakness, which can impair ambulation, delay physiotherapy and result in accidental fall.

Recent reports suggest that saphenous nerve blockade using an adductor canal approach is a novel technique with which to provide adequate analgesia for major knee surgery. Ultrasound-guided saphenous nerve block in the adductor canal is considered a technically simple and reliable block, providing consistent success. Although traditionally used to provide anesthesia and analgesia to the foot and ankle, recent reports suggest that saphenous nerve blockade in the adductor canal may provide adequate analgesia for major knee surgery. Taking into consideration the anatomy of the adductor canal, it appears possible to target not only the saphenous nerve but also multiple branches of the femoral and obturator nerve.

However, the optimal dose of local anesthetic required to establish knee analgesia without inducing quadriceps weakness has not yet been determined. Identifying an optimal dose would allow for maximum analgesic efficacy with minimal or no motor block, while minimizing other unwanted adverse effects.

This pilot study is designed to determine the optimal dose of ropivacaine 0.5% required to initiate sensory knee analgesia for the post-operative.

ELIGIBILITY:
Inclusion Criteria:

* ASA(American Society of Anesthesiologists)physical status classification system I-III
* 18-85 years of age, inclusive
* BMI 18 - 40
* Scheduled for elective total knee replacement under spinal anesthesia or general anesthesia.

Exclusion Criteria:

* Inability or refusal to provide informed consent
* Any contraindication to regional anesthesia (allergy to local anesthetics, bleeding diathesis, coagulopathy, malignancy or infection at the site of block)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2014-08-05 (Actual); Study Completion 2014-08-05 (Actual)

PRIMARY OUTCOMES:
Tolerance to Transcutaneous Electrical Stimulation (TES) | 30 min after ropivacaine injection
  To determine the minimum effective dose of ropivacaine in the adductor canal block to initiate sensory analgesia in the knee. Complete sensory anesthesia in the knee following adductor canal block 30 minutes after ropivacaine administration.

SECONDARY OUTCOMES:
The degree of motor block following ropivacaine administration | Assessments will start at baseline before ropivacaine injection and every 5 minutes after ropivacaine injection until 45 minutes have passed or until surgery commences, whichever comes first
  Motor block will be assessed using an isometric force dynamometer
Cold sensation | 30 min after ropivacaine injection
  To determine the minimum effective dose of ropivacaine in the adductor canal block to initiate sensory analgesia in the knee. Complete sensory anesthesia in the knee following adductor canal block 30 minutes after ropivacaine administration.

OTHER OUTCOMES:
Total opioid consumption | 48 hours
  Total opioid consumption during the intraoperative phase, post-operative care unit stay, and during the first 48 hours post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Vincent WS Chan, MD, Principal Investigator — University Health Network, Toronto; Richard Brull, MD, Study Chair — University Health Network, Toronto; Ki Jinn Chin, MD, Study Chair — University Health Network, Toronto; Anahi Perlas, MD, Study Chair — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Krombach J, Gray AT. Sonography for saphenous nerve block near the adductor canal. Reg Anesth Pain Med. 2007 Jul-Aug;32(4):369-70. doi: 10.1016/j.rapm.2007.04.006. No abstract available. PMID 17720129
- [Background] Casati A, Baciarello M, Di Cianni S, Danelli G, De Marco G, Leone S, Rossi M, Fanelli G. Effects of ultrasound guidance on the minimum effective anaesthetic volume required to block the femoral nerve. Br J Anaesth. 2007 Jun;98(6):823-7. doi: 10.1093/bja/aem100. Epub 2007 May 3. PMID 17478453
- [Background] Danelli G, Ghisi D, Fanelli A, Ortu A, Moschini E, Berti M, Ziegler S, Fanelli G. The effects of ultrasound guidance and neurostimulation on the minimum effective anesthetic volume of mepivacaine 1.5% required to block the sciatic nerve using the subgluteal approach. Anesth Analg. 2009 Nov;109(5):1674-8. doi: 10.1213/ANE.0b013e3181b92372. PMID 19843807
- [Background] Davis JJ, Bond TS, Swenson JD. Adductor canal block: more than just the saphenous nerve? Reg Anesth Pain Med. 2009 Nov-Dec;34(6):618-9. doi: 10.1097/AAP.0b013e3181bfbf00. No abstract available. PMID 19901788
- [Background] Manickam B, Perlas A, Duggan E, Brull R, Chan VW, Ramlogan R. Feasibility and efficacy of ultrasound-guided block of the saphenous nerve in the adductor canal. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):578-80. doi: 10.1097/aap.0b013e3181bfbf84. PMID 19916251